CLINICAL TRIAL: NCT04711200
Title: Mesenchymal Stromal Cells Treatment in Lyell Syndrome: A Pilot Phase 1-2 Open Trial
Brief Title: LYell SYndrome MEsenchymal Stromal Cells Treatment
Acronym: LYSYME
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P150941J; 2024-516404-42-00 (EU CTIS Number)
Record Dates: First submitted 2020-11-30; First posted 2021-01-15 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Epidermal Necrolysis; Lyell Syndrome; Toxic Epidermal Necrolysis; Overlap Syndrome; Mesenchymal Stromal Cells; Adipose Derived Stromal Cells
Keywords: Epidermal necrolysis; Lyell syndrome; toxic epidermal necrolysis; Overlap syndrome; Mesenchymal stromal cells; Adipose derived stromal cells
MeSH Terms: conditions — Stevens-Johnson Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adipose derived stromal cells intravenously injected (Experimental)
  Interventions: Drug: Adipose derived stromal cells intravenously injected

INTERVENTIONS:
Drug: Adipose derived stromal cells intravenously injected — 2×10^6/kg of Adipose derived stromal cells A single injection at D0 (performed maximum three days post-admission).

SUMMARY:
Stevens-Johnson syndrome (SJS) and toxic epidermal necrolysis (TEN) are rare severe cutaneous adverse reactions (SCARs) to drugs.

To date, no curative drug has demonstrated with a good level of evidence its ability to promote SJS and TEN healing and could contribute to earlier reepithelialisation. Mesenchymal stroma cells (MSCs) therapy represents a new therapeutic approach. eg, in patients with cardiovascular diseases, neurological diseases, renal transplantation, lung diseases as acute respiratory distress syndrome.

Recently, MSCs have been proposed in both burn wound healing with a significantly decrease of the unhealed burn area and in cutaneous radiation.

Moreover, MSCs have immunomodulation properties potentially effective in refractory acute and chronic graft versus host disease (GVHD) by improving thymic function and induction of Tregs. Indeed, MSCs are able to migrate to inflamed tissues after stimulation by pro-inflammatory cytokines and to modulate the local inflammatory reactions. MSCs have also demonstrated their ability to promote tissue remodelling, angiogenesis and immunomodulation through either differentiation or secretion of several growth factors such as VEGF, basic FGF and various cytokines.

Therefore, combining their immunomodulation effect and secretion of soluble factors involved in wound repair, MSCs might be valuable as a cell therapy strategy for promoting cutaneous healing in SJS-TEN syndrome and subsequently decrease the morbi-mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 and ≤ 75 years-old
* Admission ≤ 10 days after the index date (date of the first symptoms of the disease)
* Patient with confirmed SJS-TEN diagnosis hospitalized in the department of Dermatology or intensive care medicine
* At least 10 % of detachable-detached body surface area at any time during the first 10 days after the index date (date of the first symptoms of the disease)
* Who, after the nature of the study has been explained to them or a support person (if applicable), and prior to any protocol specific procedures being performed, have given written consent according to local regulatory requirements
* Affiliated to a social security scheme

Exclusion Criteria:

* Pregnant or breastfeeding women
* History of malignant disease within the past ten years and or presence of metastasis
* Positive serology for HIV
* Active infection for hepatitis B or C
* Detection of Coronavirus SARS CoV-2 RNA on admission (positive RT-PCR), if performed in the usual care
* Decompensated cardiac failure
* Uncontrolled epilepsia
* Previous history of allogenic bone marrow transplantation
* Participation in other interventional drug research Patient deprived of liberty by a judicial or administrative decision or under the protection of justice
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the research protocol and follow-up schedule
* Patient under tutorship or curatorship
* Patient under psychiatric care according to art. L1121-6 CSP

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety : Observation of at least one adverse effect | Day 10
Efficacy : Rate of complete or almost complete reepithelialisation | Day 7 after infusion

SECONDARY OUTCOMES:
Rate of observed and predicted death by the SCORTEN | at one month
Duration of hospitalisation according to our historical cohort related to BSA involved | Month 12
Duration of hospitalisation according to our historical cohort related to onset of the disease | Month 12
Duration of hospitalisation according to our historical cohort related to SCORTEN | Month 12
Duration of each mucous membranes healing ie.(buccal, nasal, genital, eyes) | at Month 12
Rate of sepsis | at Month 12
Rate of intensive care transfer | at Month 12
Rate of sequelae | at Month 12
Th1/Th2 immune response in the peripheral blood of the patients | after injection at Day 0, Day 10, Month 1
Evaluation of expression profile of Th1/Th2 associated chemokines and anti-inflammatory chemokines in the peripheral blood | after injection at Day 0, Day 10, Month 1.
Epidermal chimerism study on healed skin biopsy | at 1 month
Cutaneous re-epithelialization rate at D5, D10 and D15 post-infusion according to the percentage of cutaneous BSA re-epithelialized in comparison to maximal cutaneous detachable-detached BSA observed. | at Day 5, Day 10 and Day15

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Oro, PhD, Principal Investigator — saskia.oro@aphp.fr
Locations (1):
- Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duong TA, Valeyrie-Allanore L, Wolkenstein P, Chosidow O. Severe cutaneous adverse reactions to drugs. Lancet. 2017 Oct 28;390(10106):1996-2011. doi: 10.1016/S0140-6736(16)30378-6. Epub 2017 May 2. PMID 28476287
- [Background] Mockenhaupt M, Viboud C, Dunant A, Naldi L, Halevy S, Bouwes Bavinck JN, Sidoroff A, Schneck J, Roujeau JC, Flahault A. Stevens-Johnson syndrome and toxic epidermal necrolysis: assessment of medication risks with emphasis on recently marketed drugs. The EuroSCAR-study. J Invest Dermatol. 2008 Jan;128(1):35-44. doi: 10.1038/sj.jid.5701033. Epub 2007 Sep 6. PMID 17805350
- [Background] Creamer D, Walsh SA, Dziewulski P, Exton LS, Lee HY, Dart JK, Setterfield J, Bunker CB, Ardern-Jones MR, Watson KM, Wong GA, Philippidou M, Vercueil A, Martin RV, Williams G, Shah M, Brown D, Williams P, Mohd Mustapa MF, Smith CH. U.K. guidelines for the management of Stevens-Johnson syndrome/toxic epidermal necrolysis in adults 2016. Br J Dermatol. 2016 Jun;174(6):1194-227. doi: 10.1111/bjd.14530. No abstract available. PMID 27317286
- [Background] Roux S, Leotot J, Chevallier N, Bierling P, Rouard H. [Mesenchymal stromal cells: Biological properties and clinical prospects]. Transfus Clin Biol. 2011 Feb;18(1):1-12. doi: 10.1016/j.tracli.2011.01.001. Epub 2011 Mar 1. French. PMID 21367635
- [Background] Chung HM, Won CH, Sung JH. Responses of adipose-derived stem cells during hypoxia: enhanced skin-regenerative potential. Expert Opin Biol Ther. 2009 Dec;9(12):1499-508. doi: 10.1517/14712590903307362. PMID 19780713